CLINICAL TRIAL: NCT00002559
Title: PHASE I/II TRIAL OF TAXOL, IFOSFAMIDE, AND CISPLATIN FOR CISPLATIN-RESISTANT GERM CELL TUMOR PATIENTS WITH FAVORABLE PROGNOSTIC FEATURES
Brief Title: Combination Chemotherapy in Treating Patients With Germ Cell Tumors That Have Not Responded to Previous Cisplatin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 94-012; CDR0000063452 (Registry Identifier: PDQ (Physician Data Query)); NCI-V94-0408
Record Dates: First submitted 1999-11-01; First posted 2003-09-18 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; recurrent ovarian germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Filgrastim; Cisplatin; Ifosfamide; Paclitaxel

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: ifosfamide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy consisting of paclitaxel, cisplatin, and ifosfamide in treating patients who have ovarian or testicular germ cell tumors that are refractory to platinum-containing chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and optimal dose of paclitaxel when combined with cisplatin and ifosfamide in patients with germ cell tumors with favorable prognostic features and resistance to cisplatin.
* Determine the efficacy of this regimen as salvage therapy in these patients.

OUTLINE: This is a dose escalation study of paclitaxel.

Patients receive paclitaxel IV continuously on day 1 and cisplatin IV over 20 minutes and ifosfamide IV over 30 minutes on days 2-6. Filgrastim (G-CSF) is administered subcutaneously (SC) on days 7-18 or until blood counts recover. Treatment continues every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 3 of 6 patients experience dose-limiting toxicity. Additional patients receive paclitaxel at the MTD.

After completion of chemotherapy, some patients may undergo resection of residual masses.

PROJECTED ACCRUAL: A total of 18-43 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven germ cell tumor that is resistant to a platinum-based chemotherapy regimen
* Active disease meeting 1 of the following conditions:

  * Measurable or evaluable disease
  * Elevated serum tumor markers (alpha-fetoprotein or human chorionic gonadotropin)
  * Unresectable residual disease after postchemotherapy surgery
* Favorable prognostic factors for achieving a complete response (CR) to cisplatin-based salvage therapy required, including all of the following:

  * No more than 1 prior regimen or 6 prior courses of cisplatin
  * Testis or ovarian germ cell primary site
  * Prior CR to cisplatin therapy
  * Incomplete response to first-line therapy that was based on either carboplatin or a suboptimal regimen of cisplatin

PATIENT CHARACTERISTICS:

Age:

* 15 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8.0 g/dL

Hepatic:

* Not specified

Renal:

* Creatinine clearance greater than 50 mL/min
* Renal dysfunction due to ureteral obstruction by tumor allowed at the discretion of the principal investigator

Cardiovascular:

* If history of significant cardiac disease, evaluation and clearance by a cardiologist required prior to entry

Other:

* No active infection not well controlled on antibiotics

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No prior paclitaxel or ifosfamide
* At least 3 weeks since prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics
* Recovered from recent surgery

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 1994-01; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States